CLINICAL TRIAL: NCT05566119
Title: L5-S1 Disc Fate in Thoracolumbar Arthrodesis Stopping at L5
Acronym: L5S1OTLSF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: L5S1OTLSF
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Spinal Deformity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal deformity in adults is one of the most frequently treated pathologies in spinal surgery. Their surgical treatment remains a challenge. In particular, the choice of the borderline vertebrae for thoracolumbar fusion correction remains controversial, including the choice between an instrumented last vertebra at L5 and an arthrodesis extending to the pelvis. Studies and meta-analyses show that an ilio-sacral socket provides better correction of pelvic parameters and avoids the development of distal junctional syndrome. On the other hand, there is more proximal junctional syndrome in patients fixed to the sacrum, and the sacral socket exposes patients to the risk of pseudarthrosis of the L5-S1 level and failure of the fixation hardware. Moreover, although this factor is not described in the studies, it would seem that an ilio-sacral socket is more stiffening. Overall, no study has shown a statistically significant difference in clinical scores between patients whose last instrumented vertebra is L5 and those with pelvic fixation.

One of the theoretical risks of an extended fixation with a proximal thoracic grasp is to observe a premature disc degeneration of the L5-S1 disc since it would be subjected to more stress. This degeneration could be the cause of distal junctional syndrome and lumbo-radiculalgia due to inflammatory disc disease and disco-radicular impingement. However, to Investigator's knowledge, no clinical study has yet investigated the medium- and long-term fate of the L5-S1 disc in patients with extended fusion correction of a thoracic vertebra to L5.

Investigator's team has sometimes favored a final instrumented vertebra at L5 when possible, i.e., when the L5-S1 disc was considered to be minimally or not degenerative and when its horizontality could be obtained after correction of the underlying curvature. Investigators therefore have a cohort of patients who have undergone this technique. The usual follow-up of these patients includes a consultation appointment every 2 to 5 years and a control MRI at a distance of more than 5 years: investigators thus have a control MRI and the clinical score of the patients.

Investigator's objective is to determine whether there is degeneration of the L5-S1 disc, using MRI imaging data, which has never been published to investigator's knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Spinal fixation extended from the thorax to L5,
* Performed between 2007 (15 years of recoil and beginning of systematic preoperative MRI) and 2017 (5 years of recoil minimum)
* French speaking patient

Exclusion Criteria:

* Neuromuscular scoliosis
* Indication of fixation for fracture of ankylosed spine (impossibility of analyzing the L5-S1 disc)
* Contraindication to the realization of an MRI except if the patient has been operated on for a complementary fixation of L5-S1 in the aftermath
* Patient under guardianship or curatorship (unless consent is provided for this purpose)
* Patient deprived of liberty
* Patients who oppose participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient whose age is ≥ 18 years, with spinal fixation extended from the thorax to L5, performed between 2007 (15 years of recoil and beginning of systematic preoperative MRI) and 2017 (5 years of recoil minimum).
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Degeneration of the L5-S1 disc assessed by the Pffirman score | Year 5
  This outcome corresponds to the appearance of L5-S1 disc degradation according to the Pffirmann score between the first MRI performed as part of the preoperative workup in the 6 months prior to surgery and the 5-year follow-up MRI. The Pfirmann classification allows grading of disc degeneration at the lumbar level on T2-weighted sagittal or STIR sequences on MRI. Grade 1 corresponds to a healthy disc and is rarely observed in adults. Grade 5 corresponds to disc collapse.

SECONDARY OUTCOMES:
Pelvic parameters | Year 5
  This outcome corresponds to the variation of pelvic parameters.
Onset of spondylolisthesis | Year 5
  This outcome corresponds to the appearance of a spondylolisthesis L5-S1.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles GUERIN, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Yao YC, Kim HJ, Bannwarth M, Smith J, Bess S, Klineberg E, Ames CP, Shaffrey CI, Burton D, Gupta M, Mundis GM, Hostin R, Schwab F, Lafage V. Lowest Instrumented Vertebra Selection to S1 or Ilium Versus L4 or L5 in Adult Spinal Deformity: Factors for Consideration in 349 Patients With a Mean 46-Month Follow-Up. Global Spine J. 2023 May;13(4):932-939. doi: 10.1177/21925682211009178. Epub 2021 Apr 28. PMID 33906457
- [Background] Taneichi H, Inami S, Moridaira H, Takeuchi D, Sorimachi T, Ueda H, Aoki H, Iimura T. Can we stop the long fusion at L5 for selected adult spinal deformity patients with less severe disability and less complex deformity? Clin Neurol Neurosurg. 2020 Jul;194:105917. doi: 10.1016/j.clineuro.2020.105917. Epub 2020 May 19. PMID 32454414
- [Background] Sardar ZM, Ouellet JA, Fischer DJ, Skelly AC. Outcomes in adult scoliosis patients who undergo spinal fusion stopping at L5 compared with extension to the sacrum. Evid Based Spine Care J. 2013 Oct;4(2):96-104. doi: 10.1055/s-0033-1357360. PMID 24436707
- [Background] Jia F, Wang G, Liu X, Li T, Sun J. Comparison of long fusion terminating at L5 versus the sacrum in treating adult spinal deformity: a meta-analysis. Eur Spine J. 2020 Jan;29(1):24-35. doi: 10.1007/s00586-019-06187-8. Epub 2019 Oct 17. PMID 31624908